CLINICAL TRIAL: NCT01023360
Title: Evaluation of Antiplatelet Drug Resistance in Taiwanese With VASP & Platelet Mapping™ Assay
Brief Title: Evaluation of Antiplatelet Drug Resistance in Taiwanese With VASP & Platelet Mapping ™ Assay
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Haemonetics Corporation (Industry)
Responsible Party: Chiang Fu-Tien, PhD, National Taiwan University Hospital
Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 200804034R
Record Dates: First submitted 2008-08-07; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2008-06

CONDITIONS: 30 Healthy People
MeSH Terms: interventions — Clopidogrel; Proton Pump Inhibitors; Rabeprazole; Pantoprazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clopidogrel and proton pump inhibitors (Experimental): all participating healthy people should receive clopidogrel and 3 kinds of PPI sequentially with one week interval between each PPI.
  Interventions: Drug: Clopidogrel and proton pump inhibitors

INTERVENTIONS:
Drug: Clopidogrel and proton pump inhibitors — baseline detection --> clopidogrel 75 mg PO QD for 1 week --> clopidogrel 75 mg plus rabeprazole 20mg PO QD for 1 week --> clopidogrel 75 mg PO QD for 1 week (wash-out phase) --> clopidogrel 75 mg plus pantoprazole 40mg PO QD for 1 week --> clopidogrel 75 mg PO QD for 1 week (wash-out phase) --> clopidogrel 75 mg plus esomeprazole 40mg PO QD for 1 week -->
  1 week washout --> aspirin 100mg PO QD for 1 week
  Other Names: clopidogrel; rabeprazole; pantoprazole; esomeprazole

SUMMARY:
Currently, drugs commonly used for antiplatelet are aspirin and clopidogrel when encountering stroke or coronary heart disease. In this study, we would use VASP assay and thromboelastograph with platelet mapping assay kit to evaluate the antiplatelet resistance in general population and the relationship between clopidogrel and proton pump inhibitor.

DETAILED DESCRIPTION:
This study intent is to search the standard to diagnose of the antiplatelet drug resistance and to discover the prevalence of drug resistance in Taiwanese population in Taiwan. The trial will enroll at least 30 healthy people after fulfilling the investigation questionnaire. All the participants will receive antiplatelet drugs in two separate period and measured the efficacy by VASP assay and thromboelastograph with platelet mapping assay. The health volunteer will receive clopidogrel and different types of proton pump inhibitor to see the interference of antiplatelet efficacy between each drug.

ELIGIBILITY:
Inclusion Criteria:

* 30 Healthy people, without major systemic disease, not under medication treatment

Exclusion Criteria:

* Systemic disease, under medication control with NSAID, anticoagulants, taking antiplatelet drugs before entering trial, Chinese herb, pregnant or breast feeding woman

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of the antiplatelet drug response apparently shown in TEG & Platelet mapping assay | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tien Chiang, MD, Phd, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan